CLINICAL TRIAL: NCT02110940
Title: The Effect of Neural Mobilization Exercise on Lower Limb Pain in Patients With Rheumatoid Arthritis.
Brief Title: The Effect of Neurodynamic Mobilization Exercise on Lower Limb Pain in Patients With Rheumatoid Arthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LO CHI NGAI, Mr., The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20140401001
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative Physiotherapy (Active Comparator): Subjects will be referred to the physiotherapy department to receive conventional physiotherapy treatment.
  Interventions: Other: Conservative Physiotherapy
- Neurodynamic mobilization exercise (Experimental): The experimental group will be given three neurodynamic mobilization exercises which focus more on lower limbs and the major innervating cutaneous nerves - saphenous nerve, sciatica nerve and femoral nerve.
  Subjects will be instructed to practice everyday, each action repeat for 10 times.
  Interventions: Other: Neurodynamic mobilization exercise

INTERVENTIONS:
Other: Neurodynamic mobilization exercise — The mobilization exercise is conducted with 10 repetitions for each action, the action is hold for 5 seconds when subjects had the stretch feeling. The series of exercise is told to perform 2 sets a day, daily practice.
  Subjects' conditions will be reviewed at the end of 4th and 8th week. An exercise log book will be provided for each subject to record down the compliance of the exercise.
  Arms: Neurodynamic mobilization exercise
Other: Conservative Physiotherapy — The control group is assigned to received conventional treatment in the physiotherapy department with the standard rehabilitation protocol consisted of electrotherapy for pain relief, strengthening exercise to increase the strength of the thigh
  Arms: Conservative Physiotherapy

SUMMARY:
This clinical trial is the first study to apply neurodynamic mobilization, a nervous system specific therapeutic exercise, on patients with rheumatoid arthritis(RA). Objective of the study is to find out the effect of neurodynamic mobilization for joint inflammation in patients with RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic autoimmune disorder characterized by generalized joints inflammation. With increasing investigation on the pathology, the treatment focus on the conditions shifted from a musculoskeletal point of view to a systemic approach. The awareness of holistic treatment was also increased.

Latest studies have found out the neurogenic inflammatory mechanism played an important role in the inflammatory process of RA, the pathological changes of neural tissues in RA were also noted.

This clinical trial is the first study to apply neurodynamic mobilization, a nervous system specific therapeutic exercise, on patients with RA. Objective of the study is to find out the effect of neurodynamic mobilization for joint inflammation in patients with RA.

Population Adults who are diagnosed with Rheumatoid Arthritis.

Intervention Neurodynamic Exercise

Comparison Standard conservative physiotherapy protocol

Outcome Rheumatoid Arthritis Pain Scale (RAPS) C-reactive protein (CRP) test

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria was considered as patients with rheumatoid arthritis; presence of inflammatory condition on the joints on upper and / or lower limbs; Rheumatoid Arthritis Pain Scale (RAPS) at least 10 points during activities of daily living; and adults (> 18 years of age) in either gender.

Exclusion Criteria:

* The exclusion criteria are: acute joint pain, physiotherapy or joint injections in the previous 3 months; change in corticosteroids in the previous month; and change in disease-modifying antirheumatic drugs in the previous 3 months; subjects with poor balance or significant pain which neurodynamic mobilization is unable to perform.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Rheumatoid Arthritis Pain Scale (RAPS) | 8 weeks
  Rheumatoid Arthritis Pain Scale (RAPS) will be used to rate the severity of the pain in subjects with RA; before, between and after the experimental period. The questionnaire consists of 24 items with a scale from 0-6 to quantify the severity of the Rheumatoid Arthritis
  The test will be conducted in the baseline, at 4th week, and the end of the investigation at 8th week.

SECONDARY OUTCOMES:
C-reactive protein (CRP) test | 8 weeks
  C-reactive protein (CRP) is one of the most widely used measurements to indicate the severity of inflammation in rheumatoid arthritis. The choice of CRP is due to its cost effectiveness, reliability and reproducibility.
  The test will be coducted by nurses, a 3cc blood sample will be taken from the subject and sent to the laboratory to investigate the C-reactive protein level. The test will be conducted in the baseline, at 4th week, and the end of the investigation at 8th week.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Ngai Lo, Master, Principal Investigator
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No